CLINICAL TRIAL: NCT02627248
Title: Neoadjuvant Chemotherapy With or Without Huaier Granule in Treating Women With Locally Advanced Breast Cancer That Can Be Removed By Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Qifeng Yang, Professor, Shandong University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HECT002
Record Dates: First submitted 2015-12-03; First posted 2015-12-10 (Estimated); Last update posted 2015-12-10 (Estimated); Status verified 2015-12

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Epirubicin; Docetaxel; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Docetaxel, Epirubicin and Cyclophosphamide (TEC) (Experimental): Six cycles of docetaxel (75 mg/m²), epirubicin (70 mg/m²) and cyclophosphamide (600 mg/m²). Patients will be treated with chemotherapy every 3 weeks (+/- 2 days ) in total. Huaier Granule will be not be administrated.
  Interventions: Drug: Epirubicin; Drug: Docetaxel; Drug: Cyclophosphamide
- Docetaxel, Epirubicin and Cyclophosphamide + Huaier (TEC+HE) (Experimental): Six cycles of docetaxel (75 mg/m²), epirubicin (70 mg/m²) and cyclophosphamide (600 mg/m²). Patients will be treated with chemotherapy every 3 weeks (+/- 2 days ) in total. Huaier Granule will be administrated from the first cycle of chemotherapy until time of definitive surgery.
  Interventions: Drug: Huaier Granule; Drug: Epirubicin; Drug: Docetaxel; Drug: Cyclophosphamide
- Epirubicin and Docetaxel (ET) (Experimental): Six cycles of epirubicin (70 mg/m²) and docetaxel (75 mg/m²). Patients will be treated with chemotherapy every 3 weeks (+/- 2 days ) in total. Huaier Granule will be not be administrated.
  Interventions: Drug: Epirubicin; Drug: Docetaxel
- Epirubicin and Docetaxel+Huaier (ET+HE) (Experimental): Six cycles of epirubicin (70 mg/m²) and docetaxel (75 mg/m²). Patients will be treated with chemotherapy every 3 weeks (+/- 2 days ) in total. Huaier Granule will be administrated from the first cycle of chemotherapy until time of definitive surgery.
  Interventions: Drug: Huaier Granule; Drug: Epirubicin; Drug: Docetaxel

INTERVENTIONS:
Drug: Huaier Granule — 20g tid, orally
  Arms: Docetaxel, Epirubicin and Cyclophosphamide + Huaier (TEC+HE); Epirubicin and Docetaxel+Huaier (ET+HE)
Drug: Epirubicin — 70 mg/m² ivdrip, d1 for both TEC and ET regimes
Drug: Docetaxel — 75 mg/m² ivdrip, d2 for both TEC and ET regimes
Drug: Cyclophosphamide — 600 mg/m² ivdrip, d2 for TEC regimes
  Arms: Docetaxel, Epirubicin and Cyclophosphamide (TEC); Docetaxel, Epirubicin and Cyclophosphamide + Huaier (TEC+HE)

SUMMARY:
RATIONALE:

Huaier (Trametes robiniophila Murr) is a traditional Chinese medicine, which has been widely used in China for many years. The investigators have found that Huaier could exert synergistic effects with Epirubicin, Cyclophosphamide, and Paclitaxel on breast cancer cells. It is not yet known whether combination chemotherapy is more effective when given together with Huaier in the neoadjuvant setting .

PURPOSE:

To evaluate the effects of treatment with Huaier Granule in managing locally advanced breast cancers with synergistic action of the neoadjuvant chemotherapy.

ELIGIBILITY:
* Inclusion Criteria:

  * Age: ≥ 18, female;
  * Breast cancer (TNM II, III, IV) larger than 2cm in maximal diameter able to benefit from neoadjuvant chemotherapy;
  * Ductal or lobular histological type of the breast tumor;
  * The diagnosis and breast cancer has been confirmed by pathological examination;
  * The liver and kidney function satisfies the following conditions within 3 days after surgery (excluding day 3): aspartate aminotransferase (AST), glutamic-oxalacetic transaminase (ALT) < 2 upper limit of normal (ULN), total bilirubin ≤ 1.5 ULN, serum creatinine < 1.5 ULN;
  * Other laboratory tests meet the following requirements within 3 days after surgery (excluding day 3): Hb ≥ 90g/l, platelet count ≥ 100×109/L, absolute neutrophil count > 1.5×109/L;
  * The expected survival time ≥ 8 months;
  * The subjects volunteer to sign the informed consent.
* Exclusion Criteria:

  * Breast cancers of rare histological type (other than ductal and lobular);
  * Noninvasive cancer;
  * Presence of organ, bone, or skin metastases;
  * Pregnant or lactating women;
  * Those with active bleeding due to various reasons;
  * Those with HIV infection or AIDS-associated diseases;
  * Those with severe acute and chronic diseases;
  * Those with severe diabetes;
  * Those with serious infectious diseases;
  * Those who can not take drugs by oral route;
  * Drug abusers or those with psychological or mental diseases that may interfere with study compliance;
  * Conditions that are considered not suitable for this study investigators

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2015-10; Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Pathologic complete response (pCR) | one month after operation
  A pCR in the breast was defined as no pathologic evidence of invasive disease (residual ductal carcinoma in situ (DCIS) or lobular carcinoma in situ (LCIS) was allowed).

SECONDARY OUTCOMES:
Clinical Complete Response (cCR) | one month after the neoadjuvant chemotherapy
  A cCR was defined as achieving either a Complete Response (CR) or a Partial Response (PR) using Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. CR was defined as the disappearance of all target lesions, and PR was defined as at least a 30% decrease in the sum of the longest diameter (LD) of target lesions taking as reference the baseline sum LD.
Disease-free survival (DFS) | up to 10 years
  DFS was defined as the date of definitive surgery until the date of recurrence, metastasis, appearance of a second primary tumor, or death from any cause, whichever occurs first, assessed up to 10 years.
Overall survival (OS) | up to 10 years
  OS was defined as the date of definitive surgery until the date of death from any cause, assessed up to 10 years.

OTHER OUTCOMES:
Heterogeneity of the HR status in core biopsy and the surgical specimen | one month after operation
  Evaluation of the HR and HER2 status with immunohistochemical (IHC) staining.
Heterogeneity of the HER2 status in core biopsy and the surgical specimen | one month after operation
  Evaluation of the HR and HER2 status with immunohistochemical (IHC) staining.
Change in serum immunomodulating cytokines | up to 1 years
  Assessment of the change in serum immunomodulating cytokines by Bio-Plex Pro Assays.
The effects of Huaier Granule on adverse events of neoadjuvant chemotherapy | up to 6 months
  The adverse events were evaluated with Common Terminology Criteria for Adverse Events (CTCAE) v4.0.
The effects of Huaier Granule on sleep quality of patients | up to 2 years
  The sleep quality was evaluated with self reported VAS scale (0-10).

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu hospital of Shandong University, Ji'nan, Shandong, China

REFERENCES:
- [Background] Wang X, Qi W, Li Y, Zhang N, Dong L, Sun M, Cun J, Zhang Y, Lv S, Yang Q. Huaier Extract Induces Autophagic Cell Death by Inhibiting the mTOR/S6K Pathway in Breast Cancer Cells. PLoS One. 2015 Jul 2;10(7):e0131771. doi: 10.1371/journal.pone.0131771. eCollection 2015. PMID 26134510
- [Background] Song X, Li Y, Zhang H, Yang Q. The anticancer effect of Huaier (Review). Oncol Rep. 2015 Jul;34(1):12-21. doi: 10.3892/or.2015.3950. Epub 2015 May 5. PMID 25955759
- [Background] Kong X, Ding X, Yang Q. Identification of multi-target effects of Huaier aqueous extract via microarray profiling in triple-negative breast cancer cells. Int J Oncol. 2015 May;46(5):2047-56. doi: 10.3892/ijo.2015.2932. Epub 2015 Mar 17. PMID 25826742
- [Background] Wang X, Zhang N, Huo Q, Sun M, Dong L, Zhang Y, Xu G, Yang Q. Huaier aqueous extract inhibits stem-like characteristics of MCF7 breast cancer cells via inactivation of hedgehog pathway. Tumour Biol. 2014 Nov;35(11):10805-13. doi: 10.1007/s13277-014-2390-2. Epub 2014 Jul 31. PMID 25077927
- [Background] Wang X, Zhang N, Huo Q, Sun M, Lv S, Yang Q. Huaier aqueous extract suppresses human breast cancer cell proliferation through inhibition of estrogen receptor alpha signaling. Int J Oncol. 2013 Jul;43(1):321-8. doi: 10.3892/ijo.2013.1947. Epub 2013 May 20. PMID 23686317
- [Background] Wang X, Zhang N, Huo Q, Yang Q. Anti-angiogenic and antitumor activities of Huaier aqueous extract. Oncol Rep. 2012 Oct;28(4):1167-75. doi: 10.3892/or.2012.1961. Epub 2012 Aug 8. PMID 22895629
- [Background] Zhang N, Kong X, Yan S, Yuan C, Yang Q. Huaier aqueous extract inhibits proliferation of breast cancer cells by inducing apoptosis. Cancer Sci. 2010 Nov;101(11):2375-83. doi: 10.1111/j.1349-7006.2010.01680.x. PMID 20718753